CLINICAL TRIAL: NCT05001841
Title: Perioperative Acute Kidney Injury in Patients With Cystic Fibrosis Undergoing Lung Transplantation: a Retrospective Analysis
Brief Title: Renal Failure Following Lung Transplantation in Cystic Fibrosis Patients
Acronym: AKI_LUTX
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Professor, Policlinico Hospital
Other Study IDs: 346_2018
Record Dates: First submitted 2021-07-24; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lung Transplantation — Double lung transplant

SUMMARY:
With this retrospective observational cohort study, we performed a longitudinal assessment of the renal function of the adult CF patients who underwent LUTX, aiming 1) to describe possible risk factors associated with perioperative AKI and 2) to describe AKI short and long term effects on clinical outcomes.

DETAILED DESCRIPTION:
This study is a retrospective analysis of prospectively collected data from medical records of all consecutive CF patients who underwent LUTX at our Institution from January 2013 to December 2018.

ELIGIBILITY:
Inclusion Criteria:

* All patients with CF who underwent LUTX during the study period were considered.

Exclusion Criteria:

* single LUTX
* re-transplantation
* missing medical records;
* age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergone LUTX at a single Institution
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 1 month
  AKI stage 1, stage 2, and stage 3 whether a 1.5-1.9 times, 2-2.9 times, and >3 times increase from the preoperative creatinine was measured, respectively. Following KIDGO criteria

SECONDARY OUTCOMES:
Survival | Until May 31 2021
  Death at follow-up

OTHER OUTCOMES:
Chronic Kidney Injury | 1 year after lung transplantation
  chronic kidney disease (CKD) at 1-year follow-up was defined according to KIDGO criteria: an eGFR between 90 to 60 mL/min/1.73 m2 was considered to be stage 2 CKD, between 30-to-59 mL/min/1.73 m2 was considered to be stage 3 CKD, between mL/min/1.73 m2 was classified as stage 4, and < 15 mL/min/1.73 m2 (or need for dialysis or kidney transplant) was considered to be stage 5

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
On request